CLINICAL TRIAL: NCT04631653
Title: The Clinical Benefit of an Artificial Intelligence Software Implementation on Diabetic Retinopathy Screening
Brief Title: Verisee Software for Diabetic Retinopathy Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SE20294A
Record Dates: First submitted 2020-10-18; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Examine the diagnostic accuracy in referred participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verisee (Experimental): Screening diabetic retinopathy using Verisee software
  Interventions: Device: VeriSee®

INTERVENTIONS:
Device: VeriSee® — Screening of diabetic retinopathy using a validated deep learning-based software,VeriSee®

SUMMARY:
The investigators aim to improve the diagnostic accuracy and the clinical referral rate for diabetic retinopathy by using a deep learning-based software.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the leading cause of blindness among working-age patients with type 2 diabetes. According to previous studies, early screening and timely treatment can reduce the risk of worsening DR and blindness. International guidelines recommend that screening for DR be performed at least once every year for patients with type 2 diabetes. The investigators will implement a validated deep learning-based software, VeriSee®, in clinics, and evaluate the benefits on diagnostic accuracy and the clinical referral rate for diabetic retinopathy after implementation of this software.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients with diabetes
* Cooperation to fundal scopic examination

Exclusion Criteria:

* Diabetic duration < 5 years in patients with type 1 diabetes
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 12 months
  diagnostic accuracy compared to the baseline

SECONDARY OUTCOMES:
Screening rate of diabetic retinopathy | 12 months
  Screening rate of diabetic retinopathy in patients with diabetes
Changes in HbA1c | 3 months
  Changes in HbA1c
Referral rate of diabetic retinopathy | 12 months
  Successful referral rate for referrable diabetic retinopathy

CONTACTS AND LOCATIONS:
Overall Officials: I-Te Lee, MD,PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Division of Endocrinology and Metabolism in Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No